CLINICAL TRIAL: NCT01049880
Title: A Phase I Trial of Ascorbic Acid and Gemcitabine for the Treatment of Metastatic Pancreatic Cancer
Brief Title: A Research Trial of High Dose Vitamin C and Chemotherapy for Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Joseph J. Cullen (Other)
Collaborators: University of Iowa (Other); Holden Comprehensive Cancer Center (Other)
Responsible Party: Sponsor-Investigator, Joseph J. Cullen, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200804753
Record Dates: First submitted 2010-01-14; First posted 2010-01-15 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Pancreatic Neoplasms
Keywords: Ascorbic Acid; Gemcitabine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ascorbate (Experimental)
  Interventions: Drug: Gemcitabine with escalating ascorbic acid

INTERVENTIONS:
Drug: Gemcitabine with escalating ascorbic acid — Gemcitabine (1000 mg/m2) weekly for three weeks and then one week off. Ascorbic acid, given twice weekly, escalating doses weekly. Week 1: 15 grams ascorbic acid per infusion Week 2: 25 grams ascorbic acid per infusion Week 3: 50 grams ascorbic acid per infusion Week 4: 75 grams ascorbic acid per infusion Week 5: 100 grams ascorbic acid per infusion
  Ascorbic acid infusion dose is maintained at the level that provides a serum level of 350-400 mg/dL.
  Other Names: Gemzar; Ascor L 500

SUMMARY:
This study is designed to determine the maximum tolerated dose of vitamin C when given with a standard chemotherapy for people who have metastatic pancreatic cancer.

DETAILED DESCRIPTION:
This is a phase I, dose-escalating study of ascorbic acid (vitamin C) designed to determine the maximum tolerated dose of vitamin C or, if well tolerated, the dose required to obtain a desired ascorbic acid plasma concentration.

Because this is a phase I study, prospective subjects should have advanced disease (i.e., metastasis) and have failed other curative therapies (or, are unable to receive curative therapies due to comorbidities or stage of disease).

ELIGIBILITY:
Inclusion Criteria:

* Normal G6PD status
* Histologically or cytologically diagnosed pancreatic adenocarcinoma.
* Disease extent documented by CT scan (radiologically measurable disease is not required)
* Ambulatory patient without evidence of spinal cord compression
* No prior chemotherapy for metastatic disease
* Failed curative therapy or patient ineligible for definitive curative therapy
* Completed adjuvant therapy at least 4 weeks prior and recovered from any/all toxicities related to that treatment.
* If post-therapy, must have disease progression since that treatment
* If treated with prior radiation therapy, disease must be outside of the radiation fields
* No currently active second malignancies unless it is a non-melanoma skin cancer
* Women must be non-pregnant and non-lactating
* ECOG performance of 0, 1, or 2
* Granulocytes at least 1,500 / ul
* Platelets at least 100,000 / ul
* Creatinine less than 1.5 mg/dL or clearance of at least 60 mL / min
* Total bilirubin less than 2 times the upper limit of normal
* AST and ALT less than 3 times the upper limit of normal if liver metastases are not present. If liver metastases are present, AST and ALT less than 5 times the upper limit of normal
* PT INR less than 1.5 (unless the patient is on full dose warfarin)
* Patient must be at least 18 years of age
* Patient must be able to understand consent process, the research study, and be able to sign the consent document

Exclusion Criteria:

* A psychiatric disorder by history or examination that would prevent completion of the study
* ECOG performance of 3 or 4
* Co-morbid conditions that affect survival: end stage congestive heart failure, unstable angina, myocardial infarction (within the past 6 weeks), uncontrolled blood sugars of greater than 300 mg/dL, known chronic active hepatitis or cirrhosis.
* Consumption of excess alcohol (more than 4 drinks per day) or use of illicit drugs
* Continued sse of over-the-counter antioxidants (supplements like vitamin C and grape seeds)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-12; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Blood cell counts (neutropenia, thrombocytopenia) and serum chemistries (liver function tests, creatinine) | weekly

SECONDARY OUTCOMES:
Plasma ascorbate level (targeted to 350 to 400 mg/dL) | Weekly
Survival | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Joseph J Cullen, M.D., Principal Investigator — University of Iowa
Locations (1):
- The University of Iowa Hospitals & Clinics, Iowa City, Iowa, United States

REFERENCES:
- [Result] Welsh JL, Wagner BA, van't Erve TJ, Zehr PS, Berg DJ, Halfdanarson TR, Yee NS, Bodeker KL, Du J, Roberts LJ 2nd, Drisko J, Levine M, Buettner GR, Cullen JJ. Pharmacological ascorbate with gemcitabine for the control of metastatic and node-positive pancreatic cancer (PACMAN): results from a phase I clinical trial. Cancer Chemother Pharmacol. 2013 Mar;71(3):765-75. doi: 10.1007/s00280-013-2070-8. Epub 2013 Feb 5. PMID 23381814
- See also: Study results, free article. — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3587047/